CLINICAL TRIAL: NCT01309529
Title: Day Zero Urinary Catheter Removal in General Thoracic Surgery Patients Receiving Thoracic Epidural Analgesia: Recatheterization Rates and Urinary Tract Infection Occurrences
Brief Title: Day Zero Urinary Catheter Removal in Gen Thoracic Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Memorial Health System (Other)
Responsible Party: Laurel Rhyne, MSN, MEd, ACNP-BC, Memorial Hospital-Thoracic Program
Other Study IDs: IRB11.03.01
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Postoperative Retention of Urine; Postoperative Urinary Tract Infection
Keywords: general thoracic surgery; epidural analgesia; postoperative retention of urine; postoperative urinary tract infection; catheter associated urinary tract infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- thoracic surg, epidural, urine retention

SUMMARY:
Current standard of practice in study institution dictates day of surgery urinary catheter removal in general thoracic surgery patients receiving thoracic epidural analgesia. The investigators hypothesize that this practice results in low recatheterization rates secondary to urinary retention and low urinary tract infection rates.

DETAILED DESCRIPTION:
Study Design A prospective study design will be utilized as data will be collected in a prospective manner and standard of care/current practice will be unaltered in the patient population.

Sampling will include all patients that meet the eligibility criteria from March 01, 2011 until August 01, 2011 with a goal of forty-five patients.

Data Collection Protocol

1. The patient will be interviewed and given information regarding participation in the study by Principal Investigator and/or research team prior to surgery. Informed Consent Forms will be collected by Principal Investigator and/or research team. Principal Investigator and/or research team will collect all data on Data Collection Sheet.
2. Thoracic epidural will be placed by the anesthesiologist in pre-op per standard protocol.

   * Location of epidural will be documented by Principal Investigator and/or research team on Data Collection Sheet. (See Appendix 1)
3. Prior to surgery, if indicated, an indwelling urinary bladder catheter will be placed per pre-operative protocol.
4. Post-operative documentation of time, type and settings for epidural infusion will be documented on Data Collection Sheet.
5. Post-op eligible patients admitted to cardiothoracic step-down unit will be placed on the following protocol:

   * Thoracic Epidural will be managed by the anesthesia group.

     * Any change in prescription or dosing will be documented on the Data Collection Sheet.
   * If urinary catheter present, will be discontinued at midnight day of surgery, Day Zero; the time of discontinuation will be noted on the Data Collection Sheet.

     * If micturition occurs, amount and time will be documented on Data Collection Sheet.
     * If no spontaneous void by 0800 post-operative day (POD) 1, bladder scanning will be initiated.
     * If ≥ 400 cc per bladder scanner, the thoracic surgeon, surgeon's nurse or the Principal Investigator will not notified.
   * Any ordered interventions, the response and re- evaluation will be noted on Data Collection Sheet.

     * Urinary retention will be defined as > 400 cc and recatheterization (either intermittent or indwelling) will occur.
6. Data will only be collected during current surgery hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* All general thoracic surgery patients with a thoracic epidural catheter.

Exclusion Criteria:

* Men > 65 years old
* History of urologic procedure
* Known benign prostatic hyperplasia
* Admission to intensive care units
* History of urinary retention
* Foreign speaking patient
* Pregnant women and those less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General thoracic surgery patients with a thoracic epidural that meet the eligibility criteria admitted to a specific tertiary care facility starting March 1, 2011 and ending August 1, 2011.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-08 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate rates of recatheterization due to urinary retention and occurrence of urinary tract infections in a general thoracic surgery population receiving thoracic epidural analgesia. | 5 months
  The current standard of care at study institution is to remove urinary catheter on post operative day zero lowering urinary tract infection and recatheterization rates.

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Rhyne, ACNP-BC, Principal Investigator — Memorial Hospital-Thoracic Program
Locations (1):
- Memorial Hospital, Chattanooga, Tennessee, United States